CLINICAL TRIAL: NCT04929314
Title: A Systematic Interactive Communication Model to Strengthen Self-Care Regardless of Health Literacy Level
Brief Title: Communication Model to Self-Care - Regardless of Health Literacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Northern Denmark (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-000992-45
Record Dates: First submitted 2021-06-03; First posted 2021-06-18 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2020-12

CONDITIONS: Chronic Disease
Keywords: Health literacy; Nursing; Self-Care; Primary Care
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: The trial is single-blinded, as the participants are unaware of their group allocation. The community nurses will not be blinded, as they will know whether they perform the intervention or not.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group receive specialised nursing care that focuses on the interactive communication model. The nurses who deliver care to participants in the intervention group receive specific education and training in order to be able to provide nursing based on the interactive communication model and more individualised nursing based on health literacy level.
  Interventions: Behavioral: Systematic Interactive Communication Model to Strengthen Self-Care Regardless of Health Literacy Level
- Control (No Intervention): The participants in the control group receive usual care. The 98 municipalities in Denmark have a specialised role in community care and rehabilitation where nursing and practical help is carried out in the patients' own homes. Community care is usually provided at regular intervals based on a clinical evaluation of the patients' needs.

INTERVENTIONS:
Behavioral: Systematic Interactive Communication Model to Strengthen Self-Care Regardless of Health Literacy Level — The central element of the intervention is the interactive communication model. A website that contains easy-to-understand knowledge and material about various chronic diseases such as chronic obstructive pulmonary disease, diabetes, heart failure, as well as knowledge and material about wound care, compression treatment and prevention of infections has been developed. Information within each topic is given based on the interactive communication model. The idea is that community nurses should not themselves assess what characterizes an easy-to-understand level or the amount of information for each individual citizen, which seeks to ensure a systematic and uniformity in the work with self-care and more self-sufficient citizens. At the same time, the model makes it possible to take into account the individual citizen's knowledge and competencies (level of HL). Further, the nurses receive specialised education regarding HL to complement their use of the interactive communication model.
  Other Names: Communication Model to Self-Care - Regardless of Health Literacy
  Arms: Intervention

SUMMARY:
Healthcare systems all over the world are developing in a way that compels patients to become more active in the management of their own health and disease - a development that changes the role of modern patients and the skills needed to navigate the healthcare system. Demographic changes resulting in more elderly people have led to increases in the burden of chronic diseases and put pressure on increasingly scarce healthcare resources. One strategy for overcoming this burden is to reduce the utilization of healthcare resources in the secondary sector by reducing the length of stay and placing more health care services in the primary sector, thus allowing more rehabilitation actions, where the goal is to have patients take control of their own life situation and health.

This means that community nurses are compelled to strengthen citizens' ability to manage their own disease and everyday life. A focus on health literacy and its significance for everyday life with chronic disease can increase the probability of citizens' acquiring the instructions and guidance given by community nurses, and thus strengthen the ability for self-care and self-rehabilitation. In line with this, a systematic interactive communication model has been developed to help strengthen self-care for citizens with chronic diseases. For more information, see the description of the intervention above.

The study is targeted citizens, who receive community nursing. A possible benefit of participating is an improvement of quality of life in everyday life for citizens receiving community nursing. No risks related to participation in the study.

The study is run from four community nursing districts in Aalborg Municipality. The development of the intervention was initiated in september 2019, and the study is expected finalised in july 2022.

This study did not receive any specific grant from funding agencies in the public, commercial, or not-for-profit sectors.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Age > 18
* Fixed residence in Aalborg Municipality
* Receives home healthcare services for a period of more than three months
* Ability to speak, read and write Danish

Exclusion Criteria:

* Diagnosed with a severe psychiatric disease
* Diagnosed with dementia or other severe cognitive impairments
* Terminal
* Unable to understand and speak Danish
* Pregnancy
* Participation in other studies that could effect the primary outcome of this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Health-related quality of Life (Measured with the standardised European Quality of Life 5 Dimensions (EQ5D-3L) health-related quality of life questionnaire) | 6 months
  Health status

SECONDARY OUTCOMES:
Healthcare costs | 6 months
  Consumption of healthcare services in both primary and secondary sector (e.g. in- and outpatient costs, medication costs, costs from visiting general practitioners, and community care costs)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa KE Hæsum, Ph.D, Principal Investigator — University College of Northern Denmark
Locations (1):
- Aalborg Municipality, Aalborg, Denmark

REFERENCES:
- [Derived] Haesum LKE, Hejlesen OK, Udsen FW. An Interactive Communication Model for Self-Care-Regardless of Health Literacy: Protocol for a Quasi-Experimental Study. JMIR Res Protoc. 2023 Mar 31;12:e37673. doi: 10.2196/37673. PMID 37000515